CLINICAL TRIAL: NCT00474539
Title: A Phase 3, Randomized, Active-Controlled, Double-blind Trial Evaluating the Safety, Tolerability, and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With a Meningococcal C-Tetanus Toxoid Conjugate Vaccine and Other Routine Pediatric Vaccinations in Spain
Brief Title: Study Evaluating a 13-Valent Pneumococcal Conjugate Vaccine in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6096A1-3007
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-01

CONDITIONS: Vaccines, Pneumococcal
Keywords: Vaccine
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- 2 (Active Comparator)
  Interventions: Biological: 7-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — 1 dose at 2,4,6 and 15 months of age
  Arms: 1
Biological: 7-valent pneumococcal conjugate vaccine — 1 dose at 2,4,6 and 15 months of age
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate (13vPnC) vaccine compared to Prevenar (7vPnC), when given concomitantly with routine paediatric vaccinations in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month-old infants
* Available for the entire study period

Exclusion criteria:

* Previous vaccination with any vaccine before the start of the study
* Known contraindication to vaccination

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 449 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Spain: infomed@wyeth.com
Locations (11):
- Spain (11):
  - A Coruña
  - Almería
  - Barcelona
  - Madrid
  - Málaga
  - Ourense
  - Pamplona
  - Santiago de Compostela
  - Seville
  - Valencia
  - Vigo

REFERENCES:
- [Derived] Rodgers GL, Esposito S, Principi N, Gutierrez-Brito M, Diez-Domingo J, Pollard AJ, Snape MD, Martinon-Torres F, Gruber WC, Patterson S, Thompson A, Gurtman A, Paradiso P, Scott DA. Immune response to 13-valent pneumococcal conjugate vaccine with a reduced dosing schedule. Vaccine. 2013 Oct 1;31(42):4765-74. doi: 10.1016/j.vaccine.2013.08.009. Epub 2013 Aug 16. PMID 23965217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Spain from 4 July 2007 to 23 July 2007.
Pre-assignment Details: Participants were enrolled into the study according to the inclusion/exclusion criteria without a screening period.
Groups:
- 13vPnC: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with meningococcal C-tetanus toxoid conjugate vaccine (NeisVac-C) and combined diphtheria-tetanus-acellular pertussis (DTPa), hepatitis B, inactivated poliovirus, and hemophilus influenza type b (Hib) vaccine (Infanrix hexa) at the 2- and 4-month visits (infant series Dose 2) and one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at the 6-month visit (infant series dose 3). Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and combined DTPa, inactivated poliovirus, and hemophilus influenza type b (Hib) vaccine (Infanrix IPV + Hib) at the 15-month visit (toddler dose). Measles, mumps, and rubella vaccine (MMR) was administered without study vaccine at the 12-month visit.
- 7vPnC: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with meningococcal C-tetanus toxoid conjugate vaccine (NeisVac-C) and combined diphtheria-tetanus-acellular pertussis (DTPa), hepatitis B, inactivated poliovirus, and hemophilus influenza type b (Hib) vaccine (Infanrix hexa) at the 2- and 4-month visits (infant series Dose 2) and one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at the 6-month visit (infant series dose 3). Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and combined DTPa, inactivated poliovirus, and hemophilus influenza type b (Hib) vaccine (Infanrix IPV + Hib) at the 15-month visit (toddler dose). Measles, mumps, and rubella vaccine (MMR) was administered without study vaccine at the 12-month visit.
Period: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 223 (One participant was randomized to 7vPnC, but received 13vPnC.) | 226 (One participant was randomized to 7vPnC, but received 13vPnC.)
Vaccinated Dose 1 | 218 | 226
Vaccinated Dose 2 | 217 | 222
Vaccinated Dose 3 | 214 | 221
Completed | 213 | 220
Not Completed | 10 | 6
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Randomization error | 5 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 0 | 1
Period: After Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 213 | 220
Completed | 209 | 220
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 209 | 220
Completed | 208 | 220
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 219 | 225 | 444
Age Continuous [Mean (Standard Deviation); unit: months] | 2.1 (0.4) | 2.0 (0.4) | 2.1 (0.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 116 | 220
  Male | 115 | 109 | 224

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Serum Bactericidal Assay (SBA) Titer ≥ 1:8 in 13vPnC Group Relative to 7vPnC Group After the 2-dose NeisVac-C Infant Series
Description: Percentage of participants achieving a meningococcal C SBA serum antibody titer greater than or equal to (≥) 1:8 along with the corresponding 95% confidence interval (CI) are presented.
Time Frame: One month after infant series dose (at 5 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n)= number of participants with a determinate immunoglobulin G (IgG) antibody concentration to the given concomitant vaccine component.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC After Infant Series Dose 2: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Infanrix hexa at the 2- and 4-month visits (infant series Dose 2).
- 7vPnC After Infant Series Dose 2: Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and Infanrix hexa at the 2- and 4-month visits (infant series Dose 2).
Arm/Group | 13vPnC After Infant Series Dose 2 | 7vPnC After Infant Series Dose 2
Number analyzed (Participants) | 206 | 218
percentage of participants | 98.5 [95.8 to 99.7] | 99.1 [96.7 to 99.9]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series Dose 2 vs 7vPnC After Infant Series Dose 2; For Meningococcal C the difference in percentages between the two groups (13vPnC - 7vPnC) at >=1:8 titer was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for immune response induced by NeisVac-C was declared if the lowest limit of 2-sided 95% CI for the difference between the 2 groups (13vPnC - 7vPnC) greater than (>) -10%; Difference = -0.5, 95% CI [-3.3 to 2.0]

2. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions
Description: Local reactions were collected using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (Sig)(present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (Mod) (2.5 to 7.0 cm); Severe (Sev) (>7.0 cm). Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all participants who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC Dose 1: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Infanrix hexa at the 2-month visit.
- 7vPnC Dose 1: Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and Infanrix hexa at the 2-month visit.
- 13vPnC Dose 2: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Infanrix hexa at the 4-month visit.
- 7vPnC Dose 2: Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and Infanrix hexa at the 4-month visit.
- 13vPnC Dose 3: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa and at the 6-month visit.
- 7vPnC Dose 3: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa and at the 6-month visit.
- 13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Infanrix-IPV+Hib at the 15-month visit.
- 7vPnC Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with with NeisVac-C and Infanrix-IPV+Hib at the 15-month visit.
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 218 | 226 | 217 | 222 | 214 | 221 | 209 | 220
percentage of participants
  Tenderness-Any (n=199,205,182,180,170,175,164,172) | 21.1 | 18.5 | 21.4 | 16.1 | 10.6 | 14.3 | 28.7 | 26.7
  Tenderness-Sig (n=199,200,177,177,167,169,154,160) | 3.0 | 4.0 | 1.1 | 4.0 | 1.2 | 1.2 | 2.6 | 3.8
  Swelling-Any (n=196,200,182,177,171,170,169,168) | 13.3 | 14.5 | 22.0 | 14.7 | 23.4 | 20.0 | 26.6 | 18.5
  Swelling-Mild (n=196,200,182,177,171,170,166,168) | 12.2 | 13.0 | 20.3 | 13.0 | 20.5 | 17.1 | 22.9 | 16.0
  Swelling-Mod (n=196,196,177,175,166,168,156,163) | 2.6 | 2.0 | 2.3 | 2.3 | 6.6 | 6.0 | 9.0 | 5.5
  Swelling-Sev (n=196,196,177,175,166,168,152,156) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Redness-Any (n=197,199,181,180,172,172,170,169) | 15.2 | 15.1 | 23.8 | 20.0 | 26.7 | 22.7 | 30.0 | 23.1
  Redness-Mild (n=197,198,180,180,172,171,167,165) | 14.7 | 14.1 | 22.2 | 19.4 | 24.4 | 21.1 | 28.1 | 21.2
  Redness-Mod (n=196,197,178,175,166,169,157,163) | 0.5 | 1.0 | 2.2 | 1.1 | 3.6 | 3.6 | 9.6 | 6.7
  Redness-Sev (n=196,196,177,175,166,168,152,156) | 0.0 | 0.0 | 0.0 | 0.0 | 0.6 | 0.0 | 0.0 | 0.0

3. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events
Description: Systemic events (fever [Fv] ≥ 37.5 degrees Celsius [C], fever ≥ 38 C but ≤ 39 C, fever >39 C but ≤ 40 C, fever > 40 C, decreased (Decr) appetite, irritability, increased (Incr) sleep, decreased sleep, hives, use of medication (Meds) to treat symptoms (Sx), and use of medication to prevent symptoms were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all subjects who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 218 | 226 | 217 | 222 | 214 | 221 | 209 | 220
percentage of participants
  Fv ≥38°C, ≤39°C(n=201,204,181,189,172,176,156,169) | 22.9 | 19.6 | 32.6 | 41.8 | 20.9 | 29.0 | 31.4 | 34.3
  Fv >39°C, ≤40°C(n=196,196,177,176,166,168,154,156) | 1.0 | 0.5 | 1.7 | 1.1 | 3.6 | 3.0 | 4.5 | 2.6
  Fv >40°C (n=196,197,177,175,166,168,152,156) | 0.0 | 0.5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.7 | 0.0
  Decr appetite (n=204,207,189,191,178,178,163,178) | 31.4 | 35.7 | 46.6 | 44.0 | 37.1 | 36.0 | 31.9 | 41.0
  Irritability (n=202,211,192,190,179,188,171,179) | 46.5 | 49.8 | 57.3 | 60.0 | 43.0 | 39.4 | 41.5 | 53.6
  Incr sleep (n=204,206,189,187,175,174,162,165) | 38.7 | 39.3 | 39.2 | 36.4 | 21.1 | 27.0 | 16.7 | 24.8
  Decr sleep (n=196,204,183,187,175,178,162,166) | 19.4 | 27.5 | 27.3 | 27.8 | 22.9 | 25.3 | 19.8 | 18.7
  Meds-treat sx (n=205,209,193,197,175,189,165,177) | 41.0 | 44.5 | 54.4 | 57.9 | 39.4 | 42.9 | 50.3 | 46.9
  Meds-prevent sx(n=201,210,194,196,177,185,168,177) | 41.3 | 45.7 | 47.9 | 49.5 | 44.6 | 40.5 | 43.5 | 41.8

4. Primary Outcome: Geometric Mean Titers (GMT) for Meningococcal C Antibodies in as Measured by Serum Bactericidal Assay (SBA) 13vPnC Group Relative to 7vPnC Group After the 2-dose NeisVac-C Infant Series and the Toddler Dose
Time Frame: One month after infant series dose 2 (at 5 months of age) and one month after toddler dose (at 16 months of age)
Population: The evaluable 2-dose immunogenicity (per protocol) population was the primary analysis population consisting of eligible subjects who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Infanrix IPV + Hib at the 15-month visit (toddler dose). MMR was administered without study vaccine at the 12-month visit.
- 7vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and Infanrix IPV + Hib at the 15-month visit (toddler dose). MMR was administered without study vaccine at the 12-month visit.
Arm/Group | 13vPnC After Infant Series Dose 2 | 7vPnC After Infant Series Dose 2 | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 206 | 218 | 164 | 172
titer | 654.55 [557.75 to 768.16] | 757.04 [648.45 to 883.81] | 2573.06 [2176.29 to 3042.16] | 2098.12 [1779.65 to 2473.58]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series Dose 2 vs 7vPnC After Infant Series Dose 2; For Meningococcal C the GMT ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for or immune response induced by NeisVac-C was declared if the lower bound of the 2-sided, 95% CI for the GMT ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 0.86, 95% CI [0.69 to 1.08]
Statistical Analysis 2: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Meningococcal C the GMT ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 1.23, 95% CI [0.97 to 1.55]

5. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Diphtheria and Tetanus in 13vPnC Group Relative to 7vPnC Group After the 3-dose Infant Series and After the Toddler Dose
Description: Predefined antibody levels for Diphtheria (0.01 or 0.1 International units [IU]/mL) and Tetanus (0.01 or 0.1 [IU]/mL).
Time Frame: One month after infant series dose 3 (at 7 months of age) and one month after the toddler dose (at 16 months of age)
Population: The evaluable 3-dose immunogenicity (per protocol) population was the primary analysis population consisting of eligible subjects who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC After Infant Series Dose 3: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at the 6-month visit (infant series dose 3).
- 7vPnC After Infant Series Dose 3: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at the 6-month visit (infant series dose 3).
- 13vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Infanrix IPV + Hib at the 15-month visit (toddler dose).
- 7vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and Infanrix IPV + Hib at the 15-month visit (toddler dose).
Arm/Group | 13vPnC After Infant Series Dose 3 | 7vPnC After Infant Series Dose 3 | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 197 | 212 | 164 | 172
percentage of participants
  Diphtheria ≥0.10 IU/mL | 98.5 [95.6 to 99.7] | 99.1 [96.6 to 99.9] | 100.0 [97.8 to 100.0] | 100.0 [97.9 to 100.0]
  Diphtheria ≥0.01 IU/mL | 100.0 [98.1 to 100.0] | 100.0 [98.3 to 100.0] | 100.0 [97.8 to 100.0] | 100.0 [97.9 to 100.0]
  Tetanus ≥0.10 IU/mL | 96.6 [92.6 to 98.7] | 96.7 [93.0 to 98.8] | 100.0 [97.8 to 100.0] | 100.0 [97.9 to 100.0]
  Tetanus ≥0.01 IU/mL | 100.0 [97.9 to 100.0] | 100.0 [98.0 to 100.0] | 100.0 [97.8 to 100.0] | 100.0 [97.9 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For diphtheria the difference in percentage between the two groups (13vPnC - 7vPnC) at >=0.10 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lowest limit of 2-sided 95% CI for the difference between the 2 groups (13vPnC - 7vPnC) > -10%; Difference = -0.6, 95% CI [-3.5 to 2.0]
Statistical Analysis 2: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For diphtheria the difference in percentage between the two groups (13vPnC - 7vPnC) at >=0.01 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.0, 95% CI [-1.9 to 1.7]
Statistical Analysis 3: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For tetanus the difference in percentage between the two groups (13vPnC - 7vPnC) at >=0.10 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -0.2, 95% CI [-4.4 to 4.0]
Statistical Analysis 4: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For tetanus the difference in percentage between the two groups (13vPnC - 7vPnC) at >=0.01 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.0, 95% CI [-2.1 to 2.0]
Statistical Analysis 5: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Ratio = 0.0, 95% CI [-2.2 to 2.2]
Statistical Analysis 6: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 5, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Ratio = 0.0, 95% CI [-2.2 to 2.2]
Statistical Analysis 7: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 5, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Ratio = 0.0, 95% CI [-2.3 to 2.2]
Statistical Analysis 8: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 5, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Ratio = 0.0, 95% CI [-2.3 to 2.2]

6. Primary Outcome: Geometric Mean Antibody Concentrations (GMC) for Diphtheria and Tetanus in 13vPnC Group Relative to 7vPnC Group After the 3-dose Infant Series and After the Toddler Dose
Time Frame: One month after infant series dose 3 (at 7 months of age) and one month after the toddler dose (at 16 months of age)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- 7vPnC After Toddler Dose: SParticipants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and Infanrix IPV + Hib at the 15-month visit (toddler dose).
Arm/Group | 13vPnC After Infant Series Dose 3 | 7vPnC After Infant Series Dose 3 | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 197 | 212 | 164 | 172
IU/mL
  Diphtheria | 0.79 [0.69 to 0.90] | 0.92 [0.81 to 1.04] | 3.00 [2.63 to 3.41] | 3.23 [2.88 to 3.63]
  Tetanus | 1.10 [0.94 to 1.27] | 1.20 [1.04 to 1.39] | 3.29 [2.83 to 3.83] | 3.28 [2.83 to 3.79]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For diphtheria toxoid the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lower bound of the 2-sided, 95% CI for the GMC ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 0.86, 95% CI [0.72 to 1.03]
Statistical Analysis 2: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For tetanus the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.91, 95% CI [0.74 to 1.12]
Statistical Analysis 3: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For diphtheria toxoid the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.93, 95% CI [0.78 to 1.10]
Statistical Analysis 4: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For tetanus the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 1.00, 95% CI [0.81 to 1.24]

7. Primary Outcome: Percentage of Participants Achieving Antibody Level ≥ 0.35μg/mL in 13vPnC Group After the Second and the Third Dose of a 3-Dose Infant Series and After the Toddler Dose
Description: Percentages of participants achieving World Health Organization (WHO) predefined antibody threshold ≥ 0.35 μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after infant series dose 2 (at 5 months of age) and dose 3 (at 7 months of age) and one month after the toddler dose (at 16 months of age)
Population: The evaluable immunogenicity (per protocol) population was the primary analysis population consisting of eligible subjects who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC After Infant Series Dose 2 | 13vPnC After Infant Series Dose 3 | 13vPnC After Toddler Dose
Number analyzed (Participants) | 206 | 197 | 212
percentage of participants
  Common Serotypes - Serotype 4 | 92.5 [87.9 to 95.7] | 98.5 [95.7 to 99.7] | 100.0 [97.7 to 100.0]
  Common Serotypes - Serotype 6B | 27.9 [21.8 to 34.7] | 94.9 [90.9 to 97.5] | 100.0 [97.7 to 100.0]
  Common Serotypes - Serotype 9V | 89.9 [84.8 to 93.7] | 97.0 [93.5 to 98.9] | 99.3 [96.3 to 100.0]
  Common Serotypes - Serotype 14 | 91.0 [86.1 to 94.6] | 97.0 [93.6 to 98.9] | 99.4 [96.6 to 100.0]
  Common Serotypes - Serotype 18C | 88.9 [83.7 to 92.9] | 99.0 [96.4 to 99.9] | 98.8 [95.6 to 99.8]
  Common Serotypes - Serotype 19F | 100.0 [98.2 to 100.0] | 99.0 [96.4 to 99.9] | 98.7 [95.5 to 99.8]
  Common Serotypes - Serotype 23F | 55.8 [48.6 to 62.8] | 93.0 [88.5 to 96.1] | 98.1 [94.7 to 99.6]
  Additional Serotypes - Serotype 1 | 96.0 [92.2 to 98.2] | 98.5 [95.7 to 99.7] | 98.8 [95.6 to 99.8]
  Additional Serotypes - Serotype 3 | 73.8 [67.1 to 79.9] | 86.2 [80.5 to 90.7] | 93.6 [88.6 to 96.9]
  Additional Serotypes - Serotype 5 | 86.4 [80.8 to 90.8] | 96.0 [92.2 to 98.2] | 100.0 [97.6 to 100.0]
  Additional Serotypes - Serotype 6A | 80.8 [74.6 to 86.0] | 99.0 [96.4 to 99.9] | 99.4 [96.5 to 100.0]
  Additional Serotypes - Serotype 7F | 94.5 [90.3 to 97.2] | 100.0 [98.2 to 100.0] | 99.4 [96.5 to 100.0]
  Additional Serotypes - Serotype 19A | 92.9 [88.4 to 96.1] | 99.5 [97.2 to 100.0] | 100.0 [97.5 to 100.0]

8. Primary Outcome: Geometric Mean Antibody Concentration (GMC) in 13vPnC Group After the Second and the Third Dose of a 3-Dose Infant Series and After the Toddler Dose
Description: GMC as measured by enzyme-linked immunosorbent assay (ELISA) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMCs (13vPnC) were calculated for each pneumococcal serotype and timepoint, and 2-sided, 95% CI were constructed.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC After Infant Series Dose 2 | 13vPnC After Infant Series Dose 3 | 13vPnC After Toddler Dose
Number analyzed (Participants) | 206 | 197 | 212
μg/mL
  Common Serotypes - Serotype 4 | 1.55 [1.35 to 1.78] | 2.32 [2.08 to 2.60] | 3.88 [3.42 to 4.40]
  Common Serotypes - Serotype 6B | 0.21 [0.18 to 0.25] | 2.59 [2.20 to 3.05] | 12.25 [10.78 to 13.92]
  Common Serotypes - Serotype 9V | 1.15 [1.01 to 1.32] | 1.51 [1.35 to 1.68] | 2.67 [2.34 to 3.05]
  Common Serotypes - Serotype 14 | 1.94 [1.64 to 2.29] | 4.51 [3.89 to 5.22] | 9.82 [8.54 to 11.30]
  Common Serotypes - Serotype 18C | 1.30 [1.11 to 1.51] | 1.86 [1.68 to 2.07] | 2.29 [2.01 to 2.61]
  Common Serotypes - Serotype 19F | 2.98 [2.60 to 3.41] | 2.46 [2.21 to 2.74] | 6.11 [5.21 to 7.16]
  Common Serotypes - Serotype 23F | 0.40 [0.34 to 0.48] | 1.67 [1.44 to 1.94] | 3.96 [3.43 to 4.59]
  Additional Serotypes - Serotype 1 | 1.87 [1.61 to 2.16] | 2.95 [2.61 to 3.33] | 4.60 [3.94 to 5.37]
  Additional Serotypes - Serotype 3 | 0.54 [0.48 to 0.61] | 0.85 [0.76 to 0.95] | 1.04 [0.91 to 1.19]
  Additional Serotypes - Serotype 5 | 0.88 [0.77 to 1.00] | 1.83 [1.62 to 2.06] | 3.69 [3.26 to 4.18]
  Additional Serotypes - Serotype 6A | 0.81 [0.70 to 0.95] | 3.08 [2.76 to 3.44] | 7.71 [6.75 to 8.80]
  Additional Serotypes - Serotype 7F | 1.51 [1.33 to 1.71] | 3.41 [3.11 to 3.74] | 5.66 [4.90 to 6.53]
  Additional Serotypes - Serotype 19A | 1.52 [1.31 to 1.76] | 2.50 [2.27 to 2.75] | 10.21 [8.92 to 11.68]

9. Secondary Outcome: Percentage of Participants Achieving a Serum Bactericidal Assay (SBA) Titer ≥ 1:8 in 13vPnC Group Relative to 7vPnC Group After the Toddler Dose
Description: Percentage of participants achieving a meningococcal C SBA serum antibody titer ≥ 1:8 along with the corresponding 95% confidence interval (CI) are presented.
Time Frame: One month after toddler dose (at 16 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n)= number of participants with a determinate IgG antibody concentration to the given concomitant vaccine component.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with meningococcal C-tetanus toxoid conjugate vaccine (NeisVac-C) and combined diphtheria-tetanus-acellular pertussis (DTPa), hepatitis B, inactivated poliovirus, and hemophilus influenza type b (Hib) vaccine (Infanrix hexa) at the 2- and 4-month visits (infant series Dose 2) and one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at the 6-month visit (infant series dose 3). Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and combined DTPa, inactivated poliovirus, and hemophilus influenza type b (Hib) vaccine (Infanrix IPV + Hib) at the 15-month visit (toddler dose). Measles, mumps, and rubella vaccine (MMR) was administered without study vaccine at the 12-month visit.
- 7vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with meningococcal C-tetanus toxoid conjugate vaccine (NeisVac-C) and combined diphtheria-tetanus-acellular pertussis (DTPa), hepatitis B, inactivated poliovirus, and hemophilus influenza type b (Hib) vaccine (Infanrix hexa) at the 2- and 4-month visits (infant series Dose 2) and one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at the 6-month visit (infant series dose 3). Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and combined DTPa, inactivated poliovirus, and hemophilus influenza type b (Hib) vaccine (Infanrix IPV + Hib) at the 15-month visit (toddler dose). Measles, mumps, and rubella vaccine (MMR) was administered without study vaccine at the 12-month visit.
Arm/Group | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 164 | 172
percentage of participants | 100.0 [97.8 to 100.0] | 99.4 [96.80 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Meningococcal C the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥ 1:8 titer was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for immune response induced by NeisVac-C was declared if the lowest limit of 2-sided 95% CI for the difference between the 2 groups (13vPnC - 7vPnC) > -10%; Difference = 0.6, 95% CI [-1.7 to 3.2]

ADVERSE EVENTS:
Groups:
- 13vPnC Infant Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Infanrix hexa at the 2- and 4-month visits. Adverse events were collected from dose 1 to approximately one month after dose 3.
- 7vPnC Infant Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and Infanrix hexa at the 2- and 4-month visits. Adverse events were collected from dose 1 to approximately one month after dose 3.
- 13vPnC Post-Infant Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at the 6-month visit. Adverse events were collected from approximately one month after dose 3 to toddler dose.
- 7vPnC Post-Infant Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at the 6-month visit. Adverse events were collected from approximately one month after dose 3 to toddler dose.
- 13vPnC Toddler Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Infanrix-IPV+Hib at the 15-month visit. Adverse events were collected for approximately one month after toddler dose.
- 7vPnC Toddler Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with with NeisVac-C and Infanrix-IPV+Hib at the 15-month visit. Adverse events were collected for approximately one month after toddler dose.
- 13vPnC 6-Month Follow-up: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Infanrix hexa at the 2- and 4-month visits (infant series Dose 2) and one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at the 6-month visit (infant series dose 3). Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Infanrix IPV + Hib at the 15-month visit (toddler dose). MMR was administered without study vaccine at the 12-month visit. Adverse events were collected for approximately six months after last visit
- 7vPnC 6-Month Follow-up: Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and Infanrix hexa at the 2- and 4-month visits (infant series Dose 2) and one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at the 6-month visit (infant series dose 3). Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and Infanrix IPV + Hib at the 15-month visit (toddler dose). MMR was administered without study vaccine at the 12-month visit. Adverse events were collected for approximately six months after last visit
Arm/Group | 13vPnC Infant Series | 7vPnC Infant Series | 13vPnC Post-Infant Series | 7vPnC Post-Infant Series | 13vPnC Toddler Series | 7vPnC Toddler Series | 13vPnC 6-Month Follow-up | 7vPnC 6-Month Follow-up
Serious Adverse Events (participants affected / at risk) | 6/218 | 8/226 | 9/218 | 6/226 | 1/218 | 0/226 | 4/218 | 9/226
Other Adverse Events (participants affected / at risk) | 204/218 | 211/225 | 6/218 | 13/225 | 171/209 | 179/218 | 4/218 | 2/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Infant Series (N=218) | 7vPnC Infant Series (N=226) | 13vPnC Post-Infant Series (N=218) | 7vPnC Post-Infant Series (N=226) | 13vPnC Toddler Series (N=218) | 7vPnC Toddler Series (N=226) | 13vPnC 6-Month Follow-up (N=218) | 7vPnC 6-Month Follow-up (N=226)
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchospams (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coleliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Infant Series (N=218) | 7vPnC Infant Series (N=225) | 13vPnC Post-Infant Series (N=218) | 7vPnC Post-Infant Series (N=225) | 13vPnC Toddler Series (N=209) | 7vPnC Toddler Series (N=218) | 13vPnC 6-Month Follow-up (N=218) | 7vPnC 6-Month Follow-up (N=224)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thalassaemia beta (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 3 | 11 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 9 | 0 | 1 | 2 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 6 | 9 | 0 | 0 | 5 | 2 | 0 | 0
Irritability (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Developmental delay (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Milk allergy (Immune system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 21 | 27 | 0 | 1 | 9 | 6 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 23 | 24 | 1 | 2 | 5 | 4 | 0 | 0
Gastroenteritis (Infections and infestations) | 19 | 15 | 0 | 0 | 7 | 3 | 0 | 0
Bronchiolitis (Infections and infestations) | 12 | 17 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 9 | 14 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 9 | 13 | 0 | 1 | 1 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 5 | 8 | 0 | 0 | 1 | 1 | 0 | 0
Otitis media (Infections and infestations) | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 4 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 5 | 5 | 0 | 1 | 0 | 5 | 0 | 0
Pharyngitis (Infections and infestations) | 4 | 2 | 0 | 0 | 5 | 3 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 3 | 0 | 0 | 1 | 4 | 0 | 0
Viral infection (Infections and infestations) | 1 | 4 | 0 | 0 | 2 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Varicella (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter intestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Herpangina (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Roseola (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lice infestation (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cow's milk intolerance (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infantile asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 6 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tenderness (any) (Skin and subcutaneous tissue disorders) | 199 | 205 | 0/0 | 0/0 | 164 | 172 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (any)=present at site of vaccination.
Tenderness (any) (Skin and subcutaneous tissue disorders) | 182 | 180 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (any)
Tenderness (any) (Skin and subcutaneous tissue disorders) | 170 | 175 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (any)
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 199 | 200 | 0/0 | 0/0 | 154 | 160 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 177 | 177 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 167 | 169 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)
Induration (any) (Skin and subcutaneous tissue disorders) | 196 | 200 | 0/0 | 0/0 | 169 | 168 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose;Induration (any)=present at site of vaccination.
Induration (any) (Skin and subcutaneous tissue disorders) | 182 | 177 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (any)
Induration (any) (Skin and subcutaneous tissue disorders) | 171 | 170 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (any)
Induration (mild) (Skin and subcutaneous tissue disorders) | 196 | 200 | 0/0 | 0/0 | 166 | 163 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (mild)=0.5 centimeters (cm) to 2.0 cm.
Induration (mild) (Skin and subcutaneous tissue disorders) | 182 | 177 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (mild)
Induration (mild) (Skin and subcutaneous tissue disorders) | 171 | 170 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (mild)
Induration (moderate) (Skin and subcutaneous tissue disorders) | 196 | 196 | 0/0 | 0/0 | 156 | 163 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (moderate)=2.5 cm to 7.0 cm.
Induration (moderate) (Skin and subcutaneous tissue disorders) | 177 | 175 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (moderate)
Induration (moderate) (Skin and subcutaneous tissue disorders) | 166 | 168 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (moderate)
Induration (severe) (Skin and subcutaneous tissue disorders) | 196 | 196 | 0/0 | 0/0 | 152 | 156 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (severe) >7.0 cm.
Induration (severe) (Skin and subcutaneous tissue disorders) | 177 | 175 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (severe)
Induration (severe) (Skin and subcutaneous tissue disorders) | 166 | 168 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (severe)
Erythema (any) (Skin and subcutaneous tissue disorders) | 197 | 199 | 0/0 | 0/0 | 170 | 169 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (any)=present at site of vaccination.
Erythema (any) (Skin and subcutaneous tissue disorders) | 181 | 180 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (any)
Erythema (any) (Skin and subcutaneous tissue disorders) | 172 | 172 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (any)
Erythema (mild) (Skin and subcutaneous tissue disorders) | 197 | 198 | 0/0 | 0/0 | 167 | 165 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (mild)=0.5 centimeters (cm) to 2.0 cm.
Erythema (mild) (Skin and subcutaneous tissue disorders) | 180 | 180 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (mild)
Erythema (mild) (Skin and subcutaneous tissue disorders) | 172 | 171 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (mild)
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 196 | 197 | 0/0 | 0/0 | 157 | 163 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (moderate)=2.5 cm to 7.0 cm.
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 178 | 175 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (moderate)
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 166 | 169 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (moderate)
Erythema (severe) (Skin and subcutaneous tissue disorders) | 196 | 196 | 0/0 | 0/0 | 152 | 156 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (severe) >7.0 cm.
Erythema (severe) (Skin and subcutaneous tissue disorders) | 177 | 175 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (severe)
Erythema (severe) (Skin and subcutaneous tissue disorders) | 166 | 168 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (severe)
Fever ≥38°C but ≤39°C (General disorders) | 201 | 204 | 0/0 | 0/0 | 156 | 169 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever ≥38°C but ≤39°C
Fever ≥38°C but ≤39°C (General disorders) | 181 | 189 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥38°C but ≤39°C
Fever ≥38°C but ≤39°C (General disorders) | 172 | 176 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥38°C but ≤39°C
Fever >39°C but ≤40°C (General disorders) | 196 | 196 | 0/0 | 0/0 | 154 | 156 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >39°C but ≤40°C
Fever >39°C but ≤40°C (General disorders) | 177 | 176 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >39°C but ≤40°C
Fever >39°C but ≤40°C (General disorders) | 166 | 168 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >39°C but ≤40°C
Fever >40°C (General disorders) | 196 | 197 | 0/0 | 0/0 | 152 | 156 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >40°C
Fever >40°C (General disorders) | 177 | 175 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >40°C
Fever >40°C (General disorders) | 166 | 168 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >40°C
Decreased appetite (General disorders) | 204 | 207 | 0/0 | 0/0 | 163 | 178 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 189 | 191 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 178 | 178 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 202 | 211 | 0/0 | 0/0 | 171 | 179 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 192 | 190 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 179 | 188 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 204 | 206 | 0/0 | 0/0 | 162 | 165 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 189 | 187 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 175 | 174 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 196 | 204 | 0/0 | 0/0 | 162 | 166 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 183 | 187 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 175 | 178 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.